CLINICAL TRIAL: NCT06208917
Title: Efficacy of Ondansetron Oral Soluble Film Combined With Dexamethasone Versus Ondansetron Intravenously Combined With Dexamethasone in Prophylaxis of Chemotherapy-induced Nausea and Vomiting in Pediatric Patients : A Multi-center, Randomized, Parallel Controlled, Non-inferior Clinical Study.
Brief Title: Ondansetron (ODF) Versus Ondansetron Intravenously for the Prevention of Chemotherapy-induced Nausea and Vomiting Compare in Children
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Yizhuo Zhang (Other)
Responsible Party: Sponsor-Investigator, Yizhuo Zhang, Clinical Professor, Sun Yat-sen University
Organization: Sun Yat-sen University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SunYat-senU-ondansetron
Record Dates: First submitted 2024-01-07; First posted 2024-01-17 (Actual); Last update posted 2024-01-17 (Actual); Status verified 2024-01

CONDITIONS: Pediatric Solid Tumor, Unspecified, Protocol Specific
MeSH Terms: interventions — Ondansetron; Injections; Dexamethasone

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- oral soluble film of ondansetron combined with dexamethasone (Experimental): Participants received the first dose of ondansetron oral soluble film (age-based adjustment) 30 minutes before chemotherapy and equal doses were given 4 hours and 8 hours after the first dose for whom younger than 12 years old while the others should be given 8h hours after the first dose.
  Ondansetron oral soluble film was administered continuously for two days after chemotherapy according to the administration regimen on the day of chemotherapy. Dexamethasone (based on body surface area) iv/po twice daily from day 1 of chemotherapy until 2 days after completion of chemotherapy.
  Interventions: Drug: Ondansetron (Oral soluble film OR injections) ,Dexamethasone
- ondansetron intravenously combined with dexamethasone (Active Comparator): Participants received the first dose of ondansetron intravenously (weight-based adjustment) 30 minutes before chemotherapy and equal doses were given 4 hours and 8 hours after the first dose.
  Ondansetron (po) was given for next continuously two days in the same dose and frequency of administration. Dexamethasone (based on body surface area) iv/po twice daily from day 1 of chemotherapy until 2 days after completion of chemotherapy.
  Interventions: Drug: Ondansetron (Oral soluble film OR injections) ,Dexamethasone

INTERVENTIONS:
Drug: Ondansetron (Oral soluble film OR injections) ,Dexamethasone — Participants will randomly assigned 1:1 to receive treatment (Oral soluble film of Ondansetron plus dexamethasone OR Ondansetron injections plus dexamethasone).
  Other Names: Ondansetron，Dexamethasone

SUMMARY:
The purpose is to evaluate the efficacy of ondansetron oral soluble film plus dexamethasone in preventing chemotherapy-induced nausea and vomiting (CINV) with MEC/HEC chemotherapy in children with solid tumor.

DETAILED DESCRIPTION:
Complete randomization was used to assign subjects to the experimental group (ondansetron oral soluble film plus dexamethasone) and the control group (ondansetron intravenously plus dexamethasone) in a ratio of 1 to 1. And a specialized software was used to generate random numbers to make a random assignment table.

Experimental:

Participants received the first dose of ondansetron oral soluble film (age-based adjustment) 30 minutes before chemotherapy and equal doses were given 4 hours and 8 hours after the first dose for whom younger than 12 years old while the others should be given 8h hours after the first dose. Ondansetron oral soluble film was administered continuously for two days after chemotherapy according to the administration regimen on the day of chemotherapy. Dexamethasone (weight based) iv/po twice daily and discontinued until 72 hours after chemotherapy.

Placebo Comparator:

Participants received the first dose of ondansetron intravenously (weight-based adjustment) 30 minutes before chemotherapy and equal doses were given 4 hours and 8 hours after the first dose. Ondansetron (po) was given for next continuously two days in the same dose and frequency of administration. Dexamethasone (weight based) iv/po twice daily and discontinued until 72 hours after chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

1. Children aged 6 months to 18 years at the time of randomization;
2. Diagnosed of solid tumor by cytological or histological examination;
3. Going to initiate MEC/HEC chemotherapy;
4. PS score ≤ 2 points;
5. predicted life expectancy ≥3 months and weight greater than 6Kg;
6. Patient's parent or guardian signs informed consent

Exclusion Criteria:

1. Has vomited in the 24 hours prior to chemotherapy initiation on Treatment Day 1 ;
2. Has a symptomatic primary or metastatic central nervous system (CNS) malignancy with nausea and/or vomiting (asymptomatic participants may participate in study) ;
3. Will be receiving stem cell rescue therapy within 14 days following administration of ondansetron ;
4. Has experienced High emetic chemotherapy within two weeks ;
5. Has received or will receive total body irradiation to the abdomen or pelvis in the week prior to Treatment Day 1 and/or during the diary reporting period (120 hours following initiation of chemotherapy) ;
6. Has had benzodiazepine, opioid or opioid like therapy initiated within 48 hours prior to study drug administration, or is expected to receive within 120 hours following initiation of chemotherapy except for single doses of midazolam, temazepam or triazolam ;
7. Has started on systemic corticosteroid therapy within 72 hours prior to study drug administration or is expected to receive a corticosteroid as part of the chemotherapy regimen ;
8. Allergic to Ondansetron and dexamethasone ;
9. Has an active infection (e.g., pneumonia), congestive heart failure, bradyarrhythmia, any uncontrolled disease (e.g., diabetic ketoacidosis, gastrointestinal obstruction) except for malignancy ;
10. Is mentally incapacitated or has a significant emotional or psychiatric disorder ;
11. Has a known history of QT prolongation or is taking any medication that is known to lead to QT prolongation ;
12. Abnormal liver function (alanine aminotransferase or aspartate aminotransferase ≥ 2 times higher than the upper bound of the normal value) or abnormal renal function (serum creatinine ≥ 2.5 times higher than the upper bound of the normal value) ;
13. Is currently taking, or has taken within 48 hours of Treatment Day 1 the following drugs with antiemetic properties: 5-hydroxytryptamine 3 (5-HT3) antagonists (e.g., ondansetron), benzamides (e.g., haloperidol), cyclizine, domperidone, herbal therapies with potential antiemetic properties, olanzapine, phenothiazines (e.g., prochlorperazine), scopolamine (this is not an exhaustive list) ;
14. Has ever participated in a previous study of ondansetron or has taken an investigational drug with the last 4 weeks ;
15. other situations in which the researchers believe that they cannot be included in the group.

Ages: 6 Months to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 376 (Estimated)
Dates: Start 2023-07-09 (Actual); Primary Completion 2026-07-01 (Estimated); Study Completion 2027-01-31 (Estimated)

PRIMARY OUTCOMES:
Complete Response Rate (CR rate) | between 0 and 24 hours after the start of chemotherapy
  The proportion of patients with complete response (CRR, defined as no vomiting and no rescue therapy administered) within the acute phase (0-24h) after starting chemotherapy.

SECONDARY OUTCOMES:
CR rate in delayed phase | >24～120 Hours Post Initiation of Chemotherapy
  Complete response rate in delayed phase
CR rate in overall phase | 0~120 Hours Post Initiation of Chemotherapy
  Complete response rate in overall phase
Complete control rate in the acute, delayed, overall phases | between 0 and 120 hours after the start of chemotherapy
  Complete control rate defined as no vomiting, no rescue therapy, and no slight nausea < grade 1

CONTACTS AND LOCATIONS:
Overall Officials: Yizhuo Zhang, Principal Investigator — SunYat Sen University Cancer Center
Locations (1):
- Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China